CLINICAL TRIAL: NCT04311775
Title: The Role of Video Laryngoscope in Laryngeal Mask Placement
Brief Title: Laryngeal Mask, Video Laryngoscopy
Status: Completed | Type: Observational
Sponsor: Kocaeli Derince Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Tahsin Şimşek, medical doctor, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Other Study IDs: 2019/514/150/21
Record Dates: First submitted 2020-03-10; First posted 2020-03-17 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Difficult Intubation
Keywords: laryngeal mask

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- video laryngoscopy: video laryngoscope is a camera laryngoscope system used to see the larynx with camera
  Interventions: Device: larengeal mask insertion with video laryngoscopy
- laryngoscopy: laryngoscopy is a method used to see the larynx.
  Interventions: Other: laryngeal mask insertion

INTERVENTIONS:
Device: larengeal mask insertion with video laryngoscopy — it is a method of inserting a laryngeal mask into the airway with videolaryngoscopy
  Groups: video laryngoscopy
Other: laryngeal mask insertion — laryngeal mask is a method of inserting atube into the upper airway
  Groups: laryngoscopy

SUMMARY:
LMA insertion provide an intact airway for many surgeries during general anesthesia . LMA insertion technique was defined when it was first produced by Archie Brain . Accordingly, it is recommended to advance the device to the level where resistance is felt blindly. However, placing LMA may not always be smooth and uncomplicated. Thus, gas leaks may occur and intragastric pressure increase may occur due to gastric insufflation. To overcome these difficulties, the placement of the LMA under direct vision using a laryngoscope has been described in several studies . Previous studies have shown that the reliability of the laryngeal mask can be demonstrated by the oropharyngeal cuff leak test . In addition, the classification of the image of the laryngeal structures mediated by fiberoptic imaging and vocal cords from the LMA gives us information about the availability of effective positive pressure ventilation.

DETAILED DESCRIPTION:
LMA insertion provide an intact airway for many surgeries during general anesthesia . LMA insertion technique was defined when it was first produced by Archie Brain . Accordingly, it is recommended to advance the device to the level where resistance is felt blindly. However, placing LMA may not always be smooth and uncomplicated. Thus, gas leaks may occur and intragastric pressure increase may occur due to gastric insufflation. To overcome these difficulties, the placement of the LMA under direct vision using a laryngoscope has been described in several studies . Previous studies have shown that the reliability of the laryngeal mask can be demonstrated by the oropharyngeal cuff leak test . In addition, the classification of the image of the laryngeal structures mediated by fiberoptic imaging and vocal cords from the LMA gives us information about the availability of effective positive pressure ventilation.In cases where difficulties are found in laryngeal mask placement, using direct laryngoscope or videosingoscope, placement is frequently applied in anesthesia practice. Kim GW et al investigated LMA placement with direct laryngoscope. However, there is no study investigating the effectiveness of videongoscopes. Videoingoscopes have wide viewing angles through their cameras located at the blade tips. For this reason, we think that it will be advantageous in placing a laryngeal mask.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-65 years old
* ASA1,2,3 group patients
* Patients undergoing general anesthesia Patients scheduled for elective surgery

Exclusion Criteria:

* The patient's refusal to participate in the study
* Contraindication for placement of the laryngeal mask

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ASA1,2,3 group patients to insertion of laryngeal mask
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-02-27 (Actual)

PRIMARY OUTCOMES:
The role of Videeolaryngoscope in Placement of Laryngeal Mask | the study will comlete in two month
  video laryngoscopy use in Larengeal Mask insertion, prevent complications of Larengeal mask.

CONTACTS AND LOCATIONS:
Locations (1):
- Tahsin Şimşek, Istanbul, Kartal, Turkey (Türkiye)